CLINICAL TRIAL: NCT07236281
Title: Selenium Levels in Patients With Abdominal Aortic Aneurysm
Brief Title: Selenium Levels in Patients With Abdominal Aneurysm
Status: Active, not recruiting | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: University Hospital Bratislava (Other)
Responsible Party: Principal Investigator, Alexandra Brazinova, Chair of Institute of Epidemiology, Faculty of Medicine, Comenius University
Other Study IDs: EK 1/11/2024
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Abdominal Aneurysm; Selenium Deficiency
Keywords: abdominal aortic aneurysm; selenium deficiency
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases - persons with abdominal aortic aneurysm: Persons with abdominal aortic aneurysm (AAA) of minimally 35 mm diameter, followed by vascular surgery outpatient office. AAA is verified by radiology, was not treated by surgical or endovascular intervention.
- Controls - persons without abdominal aortic aneurysm: Persons without abdominal aortic aneurysm (AAA), as confirmed by ultrasonography. Controls will be recruited from vascular surgery outpatient office, in treatment for other vascular conditions.

SUMMARY:
Retrospective study comparing the selenium level in patients with abdominal aortic aneurysm with the selenium level in patients in the control group, i.e., patients without aneurysmal changes of the abdominal aorta.

DETAILED DESCRIPTION:
Selenium (Se), incorporated into selenocysteine, is an essential component of selenoproteins. These proteins play a crucial role in vascular protection by reducing oxidative stress, regulating inflammation, supporting endothelial nitric oxide signalling, and maintaining smooth muscle cell homeostasis. Insufficient selenoprotein activity contributes to vascular dysfunction and weakening of the vessel wall.

The aim of this project is to investigate a potential association between reduced selenium levels and abdominal aortic aneurysm (AAA) of degenerative origin.

The study group will include 20 individuals with an abdominal aortic aneurysm measuring at least 35 millimeters in diameter, verified by a radiologist using standard diagnostic imaging methods (ultrasound, CT angiography, or digital subtraction angiography). The control group will comprise 20 individuals without an abdominal aortic aneurysm. Selenium blood levels will be measured in both groups, and the relationship between selenium status and the presence of AAA will be evaluated using biostatistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* cases - patients with AAA (confirmed by radiology) followed by vascular surgery outpatient office that signed informed consent. The AAA was not treated by surgery or endovascular intervention
* controls - people without AAA (confirmed by ultrasonography) followed by vascular surgery outpatient office for other vascular disease that signed informed consent

Exclusion Criteria:

* patients that had AAA treated by surgery or endovascular intervention
* persons that did not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group comprises of 40 subjects. Twenty are cases, these are patients with AAA that was confirmed by radiology. The AAA was not treated by surgery or endovascular intervention. The are followed for the AAA by vascular surgery outpatient office. Controls are twenty persons without AAA, as confirmed by ultrasonography. They are followed by vascular surgery outpatient office for other vascular diseases. Both cases and controls are taken a blood sample, in which blood selenium level is established. Odds ratio will be calculated of having low than normal blood selenium levels in cases versus controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Odds Ratio | From enrollment to 12 months after enrollment
  Odds Ratio - odds of having lower than normal selenium levels in cases compared to the same odds in controls

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No